CLINICAL TRIAL: NCT00368589
Title: A 12 Week, Randomised, Double Blind Study Evaluating the Effects of Low Dose (10mg) and High Dose (80mg) Atorvastatin on Macrophage Activity and Carotid Plaque Inflammation as Determined by Ultra Small Super-Paramagnetic Iron Oxide (USPIO) Enhanced Carotid Magnetic Resonance Imaging (MRI)
Brief Title: Effects Of Atorvastatin On Macrophage Activity And Plaque Inflammation Using Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: TMT106468
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Atherosclerotic Carotid Disease; Atheroma; Atherosclerosis
Keywords: atherosclerotic plaque; USPIO; Atheroma; thrombo-embolic stroke; magnetic resonance imaging; Ultra small Super-Paramagnetic Iron Oxide
MeSH Terms: conditions — Carotid Artery Diseases; Plaque, Atherosclerotic; Atherosclerosis | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: atorvastatin

SUMMARY:
A new way of scanning narrowing in the arteries (main blood vessels) caused by fatty deposits known as plaques has been developed. Heart attacks and strokes occur when plaques become inflamed, depending on the artery affected. Currently used clinical tests can only tell us how much the vessel is blocked by the plaque and not how inflamed (i.e. dangerous) it is. This new method of scanning using magnetic resonance imaging (MRI) and a special agent called Sinerim can identify inflamed plaques. This study will evaluate patients with plaques in their arteries in their neck at risk of strokes to see whether treatment with a cholesterol-lowering drug called atorvastatin can reduce the amount of inflammation within the artery wall within the first three months of treatment. If this effect can be measured using MRI scanning with the use of Sinerim then the results of this study will provide additional clinical validation of the use of MRI scanning combined with agents such as Sinerem®.

ELIGIBILITY:
Inclusion criteria:

* Positive Sinerem®-enhanced MRI of carotid plaque confirmed by a consultant neuroradiologist
* Must either be statin naive or have been on a stable dose of a statin(Permitted statins and total daily dose are as follows: atorvastatin =10mg, simvastatin =40mg, pravastatin =40mg, fluvastatin =80mg, rosuvastatin =10mg for =4 weeks prior to screening, with no evidence of statin intolerability.)

Exclusion criteria:

* Require continued use of non-statin lipid modifying therapies or therapy with any other lipid regulating medications
* History of statin intolerance
* History of chronic viral hepatitis or other liver dysfunction
* Renal impairment with serum creatinine >2.5 mg/dl (>221 mol/L)
* History of myopathy or inflammatory muscle disease, or 3 times more than the upper limit of normal levels of total creatinine kinase in serum
* Doppler assessment of less than 40% stenosis during screening assessment
* Allergy to dextran and iron salts
* Contraindication to MRI scanning
* Planned carotid surgery or endovascular intervention earlier than 10 weeks within the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in USPIO-enhanced MRI signal in carotid plaques at 6 weeks and 12-weeks in low and high dose atorvastatin groups (within groups' comparison).

SECONDARY OUTCOMES:
Baseline corrected changes in USPIO-enhanced MRI signal in carotid plaques.Changes from baseline in tensile stress, micro-emboli counts, soluble plasma biomarkers at 12 weeks in low and high dose atorvastatin groups.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Clezar CN, Flumignan CD, Cassola N, Nakano LC, Trevisani VF, Flumignan RL. Pharmacological interventions for asymptomatic carotid stenosis. Cochrane Database Syst Rev. 2023 Aug 4;8(8):CD013573. doi: 10.1002/14651858.CD013573.pub2. PMID 37565307
- [Derived] Tang TY, Howarth SP, Miller SR, Graves MJ, Patterson AJ, U-King-Im JM, Li ZY, Walsh SR, Brown AP, Kirkpatrick PJ, Warburton EA, Hayes PD, Varty K, Boyle JR, Gaunt ME, Zalewski A, Gillard JH. The ATHEROMA (Atorvastatin Therapy: Effects on Reduction of Macrophage Activity) Study. Evaluation using ultrasmall superparamagnetic iron oxide-enhanced magnetic resonance imaging in carotid disease. J Am Coll Cardiol. 2009 Jun 2;53(22):2039-50. doi: 10.1016/j.jacc.2009.03.018. PMID 19477353